CLINICAL TRIAL: NCT02547350
Title: Prophylactic Intravesical Chemotherapy to Prevent Bladder Tumors After Nephroureterectomy for Primary Upper Urinary Tract Urothelial Carcinomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuesong Li (Other)
Responsible Party: Sponsor-Investigator, Xuesong Li, professor, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PIC-UTUC
Record Dates: First submitted 2015-09-08; First posted 2015-09-11 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Upper Tract Urothelial Carcinoma; Bladder Recurrence
MeSH Terms: interventions — Epirubicin; pirarubicin

ARMS (3):
- Blank control (No Intervention): do not use prophylactic intravesical chemotherapy
- single intravesical instillation (Experimental): intravesical instillation within 24 hours postoperatively
  Interventions: Drug: pharmorubicin or pirarubicin
- multiple intravesical instillation (Experimental): intravesical instillation every 1 week for the first 2 months, then once a month for the rest 10 months
  Interventions: Drug: pharmorubicin or pirarubicin

INTERVENTIONS:
Drug: pharmorubicin or pirarubicin — pharmorubicin 50mg pirarubicin 30mg
  Arms: multiple intravesical instillation; single intravesical instillation

SUMMARY:
The purpose of this study is to evaluate the efficacy of prophylactic intravesical chemotherapy (different chemotherapy drugs and dosage regimen) in the prevention of bladder recurrence after nephroureterectomy for upper tract urothelial carcinoma (UTUC).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were clinically diagnosed with UTUC
2. Treated with radical nephroureterectomy

Exclusion Criteria:

1. Distant metastasis
2. Prior history of bladder or synchronous bladder cancer
3. Administration of neoadjuvant chemotherapy
4. Presence of severe complications.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-09; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
intravesical recurrence-free survival | two years after surgery

SECONDARY OUTCOMES:
cancer-specific survival | two years after surgery